CLINICAL TRIAL: NCT03535350
Title: Phase I Study of Ibrutinib With Radiation and Temozolomide in Patients With Newly Diagnosed Glioblastoma
Brief Title: Ibrutinib With Radiation and Temozolomide in Patients With Newly Diagnosed Glioblastoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE2317
Record Dates: First submitted 2018-05-14; First posted 2018-05-24 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-01

CONDITIONS: Glioblastoma
Keywords: ibrutinib; temozolomide; brain cancer
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — ibrutinib; Radiation; Temozolomide

STUDY DESIGN:
Intervention Model Description: A standard phase 1 design will be used with 3 patients treated at each dose level and monitored for treatment-related toxicities. Escalation to the next dose will proceed in the absence of dose-limiting toxicities (DLTs).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Unmethylated MGMT Glioblastoma (Experimental): Every patient gets ibrutinib + radiation over 6 weeks. Patients will undergo a 4-week break and then Ibrutinib treatment will continue until disease progression, intolerable toxicity, or death.
  Interventions: Drug: Ibrutinib; Radiation: Radiation
- Methylated MGMT Glioblastoma (Experimental): Every patient gets ibrutinib + radiation + daily Temozolomide (TMZ) (75mg/m2) for 6 weeks. Patients will undergo a 4-week break and patients will then receive daily ibrutinib and adjuvant Temozolomide for Days 1-5 of a 28-day cycle of temozolomide for 6 cycles. The temozolomide will continue until disease progression, intolerable toxicity, or death or maximum of 6 cycles. Ibrutinib treatment will continue until disease progression, intolerable toxicity, or death.
  Interventions: Drug: Ibrutinib; Radiation: Radiation; Drug: Temozolomide (TMZ)

INTERVENTIONS:
Drug: Ibrutinib — Dose response of Ibrutinib. Level 1 starting dose is 420mg daily. Level 2 starting dose is 560mg daily. Level -1 starting dose is 280mg daily.
  November 2020:
  420 mg of ibrutinib plus temozolomide and radiation was found to be safe - up to 36 participants can betreated at the expansion cohort in both arm 1 and arm 2.
  Other Names: Imbruvica
Radiation: Radiation — 2Gy x 30minutes for 6 weeks.
Drug: Temozolomide (TMZ) — Cycle 1 150mg/m2 and cycle 2-6 will be up to 200mg/m2.
  Other Names: Temodar; Methazolastone
  Arms: Methylated MGMT Glioblastoma

SUMMARY:
Safety of combination of ibrutinib and radiation at various dose levels in unmethylated o6-methylguanine-DNA-methyltransferase (MGMT) glioblastoma and study of ibrutinib, temozolomide, and radiation combination therapy in methylated MGMT glioblastoma.

DETAILED DESCRIPTION:
There are a number of brain tumor studies including those in NCI consortium that are not including temozolomide for increased toxicity with novel agents or other drugs when added to temozolomide and radiation. However, if the combination of ibrutinib and radiation in unmethylated MGMT glioblastoma patient population is safe at every dose level we can study the safety of ibrutinib, radiation and Temozolomide in the methylated patient population. Concomitant use of radiation will lead to break down of the blood brain barrier and increase ibrutinib delivery to the brain tumor and hence the rationale to combine ibrutinib with radiation with or without temozolomide.

November 2020:

420 mg of ibrutinib plus temozolomide and radiation was found to be safe - up to 36 participants can be treated at the expansion cohort in both arm 1 and arm 2.

ELIGIBILITY:
Inclusion Criteria:

Arm 1:

* Supratentorial unmethylated MGMT glioblastoma
* Gadolinium MRI or contrast CT within 28 days of starting treatment
* Karnofsky performance ≥ 70% (http://www.npcrc.org/files/news/karnofsky_performance_scale.pdf)
* Absolute neutrophil count > 1500/mm3, platelets > 100,000/mm3, Creatinine ≤ 1.7 mg/dl, total bilirubin ≤ 1.5mg/dl, transaminases ≤ 3 times above the upper limits of normal
* Must be able to provide written informed consent
* Patients of reproductive potential must use an acceptable form of birth control to avoid contraception during the period of therapy and up to 90 days after the last dose of study drug. (eg. implants, injectable, oral contraceptives, intrauterine device (IUD), abstinence, and a barrier method which includes, but is not limited to condoms, vaginal rings, and sponges)
* Female patients must have a negative pregnancy test upon study entry.
* No concurrent malignancy with the exception of curatively treated early stage bladder and prostate cancer, basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix and breast, adequately treated stage I or II cancer from which the patient is in complete remission. Any other prior malignancies must be disease free for ≥ 3 years.
* Prothrombin time (PT) / international normalized ratio (INR) < 1.5 x upper limit of normal (ULN) and partial thromboplastin time (PTT) (aPTT) < 1.5 x ULN
* Patient with any surgery more than stereotactic biopsy are eligible so that there is enough tissue for MGMT analysis.

Arm 2:

* Arm 1 inclusion criteria must be met with the exception of the histology of the cancer, which must be methylated MGMT glioblastoma

Exclusion Criteria:

* Serious concurrent infection or illness
* Patients who are pregnant or breastfeeding
* Patients receiving concurrent therapy for their tumor
* Concurrent or prior malignancy unless curatively treated carcinoma-in-situ or basal cell carcinoma of the skin.
* Repeat craniotomy for tumor therapy after receiving radiation and TMZ treatment.
* Patients who received other chemotherapy or investigational agents in addition to radiation therapy and accompanying TMZ treatment.
* Previous ibrutinib or other Bruton's tyrosine kinase (BTK) inhibitor use or allergies to components of the study drug.
* Use of anticoagulants (including warfarin, other coumadin-derivative anticoagulant, vitamin K antagonists, or low molecular weight heparin)
* Use of drugs known to be moderate and strong inhibitor or inducers of the P450 isoenzyme CYP3A. Participants must be off P450/CYP3A inhibitors and inducers for at least a week prior to starting the study drug.
* Active, significant liver impairment (Child-Pugh class B or C)
* Patient is using systemic immunosuppressant therapy, including cyclosporineA, tacrolimus, sirolimus, and other such medications, or chronic administration of > 5 mg/day or prednisone or the equivalent.Participants must be off of immunosuppressant therapy for at least 21days prior to the first dose of the study drug. Patients can be on steroids for brain edema.
* Significant EKG abnormalities and active and significant cardiovascular disease within 6 months of screening.
* Pregnant or breastfeeding women. Male patients that intend to father a child while enrolled or 90 days after the last dose of the study drug.
* Unwillingness to comply with the protocol
* Uncontrolled, active systemic infection.
* Major surgery within 4 weeks of first dose of study drug.
* Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug.
* Recent infection requiring systemic treatment that was completed ≤ 14 days before the first dose of study drug.
* Known bleeding disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-08-24 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of ibrutinib | 6 weeks
  Determination of MTD of Ibrutinib with methylated or unmethylated glioblastoma

SECONDARY OUTCOMES:
Number of patients who experience adverse events | 10 weeks
  Safety of combination of Ibrutinib with Radiation or Ibrutinib with Temozolomide and Radiation
Number of patients with Progression Free Survival (PFS) | 10 weeks
  Number of patients that are alive without disease progression
Length of time of overall survival | 10 weeks
  Patient survival at time of last assessment

CONTACTS AND LOCATIONS:
Overall Officials: David Peereboom, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States